CLINICAL TRIAL: NCT05060640
Title: PREVALENCE OF ANAL PRECANCEROUS LESIONS IN HIGH-RISK PATIENTS DETECTED BY ROUTINE COLONOSCOPY (PACCO STUDY)
Brief Title: ANAL PRECANCEROUS LESIONS IN HIGH-RISK PATIENTS.
Acronym: PACCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Fernando Pessoa (Other)
Responsible Party: Sponsor
Other Study IDs: 78A
Record Dates: First submitted 2021-09-17; First posted 2021-09-29 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: AIN3; AIN2; HSIL, High Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Detection of anal HSIL in a routine colonoscopy. — Detection of anal HSIL in a routine colonoscopy by using acetic acid and NBI/BLI.

SUMMARY:
HIV-positive patients, women with a history of genital neoplasia and patients under pharmacologically immunosuppression (e.g. transplanted recipients, Crohn´s disease and Lupus) are a high-risk population for anal human-papillomavirus infection and associated complications, like anal precancerous lesions and anal squamous cell carcinoma. There is a lack of information on the prevalence of anal precancerous detected by routine colonoscopy in this population, by evaluating the squamocolumnar junction (the most susceptible area for lesions) during this procedure. Given, the increasing incidence rates of anal squamous cell carcinoma expected for the next two decades and the increase number of at-risk patients, the possible benefit of routine endoscopy in the diagnosis of anal precancerous lesions needs to be further explored.

DETAILED DESCRIPTION:
Procedures in all patients:

1. Digital anorectal evaluation
2. Colonoscopy with retroflection and visualization of the anal squamocolumnar junction
3. After identification of this area 5% acetic acid will be applied.
4. Visualization under NBI/BLI.
5. Biopsies of all the suspected lesions of anal high-grade squamous lesions (HSIL).

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive patients
2. Solid transplanted recipients
3. Crohn's disease patients under immunosuppression: steroids, thiopurines, biologics
4. Patients with lupus under immunosuppression
5. Women with a previous history of genital neoplasia (high-grade lesions or cancer) in the cervix, vagina or vulva.

Exclusion Criteria:

1. Previous anal/perianal cancer history
2. Previous known history of anal/perianal intraepithelial neoplasia
3. Pelvic radiation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-positive patients, women with genital neoplasia (cervix, vulva and vagina), solid organ transplanted recipients, patients with inflammatory bowel disease and patients with Lupus.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of anal high-grade squamous intraepithelial lesions in the squamocolumnar junction detected during routine colonoscopy. | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Pessoa Teaching Hospital, Gondomar, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided